CLINICAL TRIAL: NCT06534450
Title: A Comparative Randomized Placebo (Sham Pheresis) Controlled Clinical Trial To Evaluate The Effects Of Therapeutic Plasma Exchange (TPE) On Age Related Biomarkers And Epigenetics
Brief Title: The Effects Of Therapeutic Plasma Exchange (TPE) On Age Related Biomarkers And Epigenetics
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dobri Kiprov (Industry)
Collaborators: CIRCULATE, Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Dobri Kiprov, Chief Medical Officer, Global Apheresis, Inc.
Organization: Global Apheresis, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 7348
Record Dates: First submitted 2024-07-17; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Aging
Keywords: Therapeutic Plasma Exchange
MeSH Terms: interventions — Plasma Exchange; Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- TPE Monthly (Active Comparator): will receive 6 monthly TPE procedures (TOTAL 6 treatments)
  Interventions: Device: Therapeutic Plasma Exchange
- TPE Bimonthly (Active Comparator): will receive 2 TPE procedures in one week. The same treatment will be repeated on a monthly basis two more times (Two treatments per month for three months to total 6 treatments)
  Interventions: Device: Therapeutic Plasma Exchange
- TPE Bimonthly with IVIG (Active Comparator): will receive 2 TPE procedures followed by 2 gm of IVIG in one week. The same treatment will be repeated on a monthly basis twice more. (Two TPE procedures per month for three months - total of 6 treatments)
  Interventions: Device: Therapeutic Plasma Exchange; Drug: IVIG
- Sham (Sham Comparator): Sham TPE PROCEDURE once a month for 6 months (total of 6 treatments)
  Interventions: Device: Sham

INTERVENTIONS:
Device: Sham — The patient's blood will not circulate through the apheresis machine. The patient will receive approximately 250 cc of normal saline during each sham pheresis procedure.
  Arms: Sham
Device: Therapeutic Plasma Exchange — Blood is withdrawn from a peripheral or central vein into the blood cell separator which separates the whole blood into plasma and cell components. The plasma is removed and the blood cells are returned to the patient along with replacement fluids, most commonly 5% human albumin in normal saline.
  Arms: TPE Bimonthly; TPE Bimonthly with IVIG; TPE Monthly
Drug: IVIG — Intravenous Immunoglobulin
  Arms: TPE Bimonthly with IVIG

SUMMARY:
The goal of this clinical trial is to assure the safety of long term therapeutic plasma exchange (TPE) with and without Intravenous Immunoglobulin (IVIG) and its effects on biomarkers and epigenetic biologic clocks in forty individuals. The main question is to assure the safety from long term TPE using changes in clinical and laboratory outcomes and also evaluating changes on additional blood biomarkers and epigenetic clocks during and after TPE treatment. Researchers will compare the TPE treatment group to the Sham treatment group to identify changes due to TPE. Participants will receive six TPE or Sham treatments over one of two treatment schedules and may receive IVIG with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 50 years of age with or without chronic inflammatory condition

Exclusion Criteria:

* Poor peripheral vascular access
* Diagnosis of active malignancy
* Late-stage Alzheimer's disease Any medical condition which may deteriorate because of plasma exchange procedures. These include, but are not limited to, symptomatic coronary artery disease, congestive heart failure and restrictive pulmonary disease (COPD). The investigators reserve the right to exclude anyone they feel may be harmed in any way by participating in the trial.
* Presence of active infection
* Alcohol or drug dependency
* Psychiatric disorder that will interfere with participation in the study (e.g., schizophrenia, bipolar disorder)

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events and unanticipated events total for TPE safety | through study completion, an average of 1 year
  The primary objective is to assure the safety of long term TPE
Rate of change to blood epigenetic clock from TPE | through study completion, an average of 1 year
  The objective is to compare the rate of change to the blood epigenetic clock from TPE.

SECONDARY OUTCOMES:
Change in hand grip strength | after study completion, an average of 2 years
  The objective is to compare changes in hand grip strength from TPE
Change in time up and go test | after study completion, an average of 2 years
  The objective is to compare changes in the time up and go test from TPE
Change in balance time | after study completion, an average of 2 years
  The objective is to compare changes in balance time from TPE
Change in short-form health survey score | after study completion, an average of 2 years
  The objective is to compare changes in short-form health survey scores from TPE, with higher scores being better

CONTACTS AND LOCATIONS:
Overall Officials: Dobri Kiprov, MD, Principal Investigator — Global Apheresis
Locations (1):
- Global Apheresis, Mill Valley, California, United States

REFERENCES:
- [Derived] Fuentealba M, Kiprov D, Schneider K, Mu WC, Kumaar PA, Kasler H, Burton JB, Watson M, Halaweh H, King CD, Yuksel ZS, Roska-Pamaong C, Schilling B, Verdin E, Furman D. Multi-Omics Analysis Reveals Biomarkers That Contribute to Biological Age Rejuvenation in Response to Single-Blinded Randomized Placebo-Controlled Therapeutic Plasma Exchange. Aging Cell. 2025 Aug;24(8):e70103. doi: 10.1111/acel.70103. Epub 2025 May 27. PMID 40424097